CLINICAL TRIAL: NCT05351216
Title: The Effect of Sirolimus on Time-sequentially Scheduled Immunizations During the Treatment of Kaposiform Hemangioendothelioma: a Case-control Study
Brief Title: The Effect of Sirolimus on Immunizations During the Treatment of Kaposiform Hemangioendothelioma
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: LK220323
Record Dates: First submitted 2022-03-30; First posted 2022-04-28 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Kaposiform Hemangioendothelioma
Keywords: Following National Vaccination Program; Sirolimus
MeSH Terms: conditions — Kaposiform Hemangioendothelioma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Individuals diagnosed with KHE and treated with sirolimus. After immunoglobulin and flow cytometry assays, as well as outpatient evaluation and assessment, those participants will be vaccinated with live attenuated vaccines or inactivated vaccines in a timely order according to the advice. （Sirolimus Rapamycin 0.8mg/m2 bid po）
- Controls: Healthy children with no immunodeficiency disease, vaccinated according to the National Immunization Program. Particpants should be age-matched with the case group.

INTERVENTIONS:
Other:  — No intervention

SUMMARY:
To research and explore the antibody protection and immune memory after vaccination in children with KHE during sirolimus administration. To explore the feasibility (safety and efficacy) of vaccination in a timely manner during the administration of sirolimus in children with KHE. To search for back-up plans for vaccination regimens for KHE patients taking sirolimus in children who do not respond to primary vaccination.

DETAILED DESCRIPTION:
Children with KHE have an early onset. KHE usually occurs in infants and young children less than 1 year old, of which neonates account for about 38.5%-60% of all cases. Due to the immunosuppressive effect of sirolimus, the vaccination was usually suspended after taking it, and children would be in a state of no immune protection. These children are at greatly increased risk of exposure to microorganisms and consequent infection. Therefore, it is necessary to vaccinate them against infectious diseases. However, vaccination with live vaccines has the potential to cause severe infections through reversion of the vaccine strain to a pathogenic form. Moreover, studies have also shown that protective antibodies are severely affected in transplant patients taking immunosuppressive drugs and in patients with solid tumors after chemotherapy. Loss of immune memory is very common, and marked deficits in B cell function and humoral immunity can persist even for years.

ELIGIBILITY:
Inclusion Criteria:

* Case groups:
* KHE patients treated with sirolimus.
* After immunoglobulin and flow cytometry assays, as well as outpatient evaluation and assessment, those participants will be vaccinated with live attenuated vaccines or inactivated vaccines in a timely order according to the advice.
* Control groups:
* Healthy children with no immune deficiencies.
* Participants are vaccinated according to the National Immunization Program in a timely manner.
* Participants are matched to the case group according to age.

Exclusion Criteria:

* HBsAg, HBeAg positive, or other active infectious diseases;
* History of immunodeficiency or low immunoglobulin levels;
* Autoimmune disease or fever during blood collection;
* Use of other medication or surgery;
* Suffering from other bleeding disorders;
* Suffering from other solid tumors or hematological tumors, etc.;
* Withdraw informed consent.

Max Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The calculation of the sample size came from the previous pre-experiment. Investigator take HBsAb protection rate as the main outcome indicator. The sample size of this study, calculated using a non-inferiority test, was 156 (78 per group). In addition, 10% was required to make up for loss to follow-up, withdrawal, etc. So a total of 174 subjects (87 per group) are anticipated.
Sampling Method: Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Titers of Hepatitis B virus surface antibody | Admission within 1 day
  Titers of Hepatitis B virus surface antibody，indicating whether there is persistent protective antibodies after vaccination.
Titers of Hepatitis B virus surface antibody | The 7th month after admission
  Titers of Hepatitis B virus surface antibody，indicating whether there is persistent
Titers of Hepatitis B virus surface antibody | The 12th month after admission
  Titers of Hepatitis B virus surface antibody，indicating whether there is persistent
Titers of Hepatitis B virus surface antibody | The 18th month after admission
  Titers of Hepatitis B virus surface antibody，indicating whether there is persistent

SECONDARY OUTCOMES:
Levels of measles antibodies. | Admission within 1 day
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Levels of mumps antibodies | Admission within 1 day
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Levels of rubella antibodies. | Admission within 1 day
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Levels of measles antibodies. | The 7th month after admission
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Levels of mumps antibodies. | The 7th month after admission
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Levels of rubella antibodies. | The 7th month after admission
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Levels of measles antibodies. | The 12th month after admission
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Levels of mumps antibodies. | The 12th month after admission
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Levels of rubella antibodies. | The 12th month after admission
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Levels of measles antibodies. | The 18th month after admission
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Levels of mumps antibodies. | The 18th month after admission
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Levels of rubella antibodies. | The 18th month after admission
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Level of Japanese encephalitis antibody. | Admission within 1 day
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Level of Japanese encephalitis antibody. | The 7th month after admission
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Level of Japanese encephalitis antibody. | The 12th month after admission
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Level of Japanese encephalitis antibody. | The 18th month after admission
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Level of varicella antibody | Admission within 1 day
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Level of varicella antibody. | The 7th month after admission
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Level of varicella antibody. | The 12th month after admission
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Level of varicella antibody. | The 18th month after admission
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Level of COVID-19 antibody. | Admission within 1 day
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Level of COVID-19 antibody. | The 7th month after admission
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Level of COVID-19 antibody. | The 12th month after admission
  This outcome indicates whether there is persistent protective antibodies after vaccination.
Level of COVID-19 antibody. | The 18th month after admission
  This outcome indicates whether there is persistent protective antibodies after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Li, PhD, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Zignol M, Peracchi M, Tridello G, Pillon M, Fregonese F, D'Elia R, Zanesco L, Cesaro S. Assessment of humoral immunity to poliomyelitis, tetanus, hepatitis B, measles, rubella, and mumps in children after chemotherapy. Cancer. 2004 Aug 1;101(3):635-41. doi: 10.1002/cncr.20384. PMID 15274078
- [Background] Kwon HJ, Lee JW, Chung NG, Cho B, Kim HK, Kang JH. Assessment of serologic immunity to diphtheria-tetanus-pertussis after treatment of Korean pediatric hematology and oncology patients. J Korean Med Sci. 2012 Jan;27(1):78-83. doi: 10.3346/jkms.2012.27.1.78. Epub 2011 Dec 19. PMID 22219618
- [Background] Zhang J, Xie F, Delzell E, Chen L, Winthrop KL, Lewis JD, Saag KG, Baddley JW, Curtis JR. Association between vaccination for herpes zoster and risk of herpes zoster infection among older patients with selected immune-mediated diseases. JAMA. 2012 Jul 4;308(1):43-9. doi: 10.1001/jama.2012.7304. PMID 22760290
- [Background] Kawano Y, Suzuki M, Kawada J, Kimura H, Kamei H, Ohnishi Y, Ono Y, Uchida H, Ogura Y, Ito Y. Effectiveness and safety of immunization with live-attenuated and inactivated vaccines for pediatric liver transplantation recipients. Vaccine. 2015 Mar 17;33(12):1440-5. doi: 10.1016/j.vaccine.2015.01.075. Epub 2015 Feb 7. PMID 25665961
- [Background] Inoue T, Moran I, Shinnakasu R, Phan TG, Kurosaki T. Generation of memory B cells and their reactivation. Immunol Rev. 2018 May;283(1):138-149. doi: 10.1111/imr.12640. PMID 29664566
- [Background] Vink P, Ramon Torrell JM, Sanchez Fructuoso A, Kim SJ, Kim SI, Zaltzman J, Ortiz F, Campistol Plana JM, Fernandez Rodriguez AM, Rebollo Rodrigo H, Campins Marti M, Perez R, Gonzalez Roncero FM, Kumar D, Chiang YJ, Doucette K, Pipeleers L, Aguera Morales ML, Rodriguez-Ferrero ML, Secchi A, McNeil SA, Campora L, Di Paolo E, El Idrissi M, Lopez-Fauqued M, Salaun B, Heineman TC, Oostvogels L; Z-041 Study Group. Immunogenicity and Safety of the Adjuvanted Recombinant Zoster Vaccine in Chronically Immunosuppressed Adults Following Renal Transplant: A Phase 3, Randomized Clinical Trial. Clin Infect Dis. 2020 Jan 2;70(2):181-190. doi: 10.1093/cid/ciz177. PMID 30843046
- [Background] Saghafian-Hedengren S, Soderstrom I, Sverremark-Ekstrom E, Nilsson A. Insights into defective serological memory after acute lymphoblastic leukaemia treatment: The role of the plasma cell survival niche, memory B-cells and gut microbiota in vaccine responses. Blood Rev. 2018 Jan;32(1):71-80. doi: 10.1016/j.blre.2017.08.009. Epub 2017 Aug 26. PMID 28886882
- [Background] Horns F, Dekker CL, Quake SR. Memory B Cell Activation, Broad Anti-influenza Antibodies, and Bystander Activation Revealed by Single-Cell Transcriptomics. Cell Rep. 2020 Jan 21;30(3):905-913.e6. doi: 10.1016/j.celrep.2019.12.063. PMID 31968262
- [Background] Dini G, Toletone A, Barberis I, Debarbieri N, Massa E, Paganino C, Bersi F, Montecucco A, Alicino C, Durando P. Persistence of protective anti-HBs antibody levels and anamnestic response to HBV booster vaccination: A cross-sectional study among healthcare students 20 years following the universal immunization campaign in Italy. Hum Vaccin Immunother. 2017 Feb;13(2):440-444. doi: 10.1080/21645515.2017.1264788. PMID 27925503
- [Background] Zhang L, Thornton CP, Ruble K, Cooper SL. Post-Chemotherapy Titer Status and Need for Revaccination After Treatment for Childhood Cancer. Clin Pediatr (Phila). 2020 Jun;59(6):606-613. doi: 10.1177/0009922820915884. PMID 32423345